CLINICAL TRIAL: NCT01466855
Title: A Pilot Study of Intra-Ophthalmic Artery Topotecan Infusion for the Treatment of Retinoblastoma
Brief Title: A Study of Intra-Ophthalmic Artery Topotecan Infusion for the Treatment of Retinoblastoma
Acronym: IARB1
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Competing studies
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IARB1
Record Dates: First submitted 2011-10-19; First posted 2011-11-08 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2017-02

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Retinoblastoma (Experimental): Study of Intra-Ophthalmic Artery Topotecan infusion for the Treatment of Retinoblastoma.
  Interventions: Drug: Intra-Ophthalmic Artery Topotecan Infusion

INTERVENTIONS:
Drug: Intra-Ophthalmic Artery Topotecan Infusion — Topotecan via intra-ophthalmic artery delivery infused over 30 minutes on Day 1 of every 21-day cycle.

SUMMARY:
This study will test if giving topotecan directly into the blood vessel of the eye will improve the treatment of retinoblastoma. This method is referred to as "selective intra-ophthalmic artery chemotherapy" (SIOAC).

The goals of this study are:

* To find out if topotecan is an effective treatment for retinoblastoma when delivered directly to the ophthalmic artery (SIOAC delivery)
* To find out what kind of effects (good and bad) can be expected when topotecan is given by SIOAC
* To assess visual pathway function before and after the study therapy
* To learn more about the pharmacology (how your body handles the drug) of topotecan when delivered directly to the ophthalmic artery

ELIGIBILITY:
Inclusion Criteria:

1. Age: 15 years of age or younger
2. Diagnosis: Patients with untreated Group C/D/E unilateral Retinoblastoma at presentation without an indication for immediate enucleation (neovascular glaucoma or orbital pain) (Stratum A), or patients with a history of bilateral retinoblastoma and recurrent and/or refractory intraocular retinoblastoma where chemotherapy, external beam radiation and/or enucleation remain the only known option for disease control (Stratum B).
3. Therapeutic Options: Chemotherapy, External Beam Radiation therapy and/or Enucleation
4. Lansky ≥ 50 for patients ≤ 10 years of age; Karnofsky ≥ 50 for patients > 10 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Prior Therapy: Stratum A: No prior therapy is allowed. Stratum B: Patients must have local relapsed/refractory disease after receiving standard upfront therapy involving at least one chemotherapeutic regimen. There is no limit to prior chemotherapeutic regimens permitted. Prior radiation therapy is permitted.
6. Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study, as described below:

   * Myelosuppressive chemotherapy: patients must not have received myelosuppressive chemotherapy within 3 weeks of study enrollment.
   * Biologic therapies: Patients must not have received biologic anti-cancer agents within one week of study enrollment.
   * Radiation therapy: Four weeks must have elapsed since external beam radiation therapy, if given.
7. Adequate Bone Marrow Function Defined as:

   * Peripheral absolute neutrophil count (ANC) greater than or equal to 750/uL
   * Platelet count greater than or equal to 75,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to enrollment)
   * Hemoglobin greater than or equal to 8.0 gm/dL (may receive RBC transfusions)
8. Adequate Renal Function Defined as:

   -Maximum serum creatinine based on age as follows: 1 to < 2 years- 0.6 mg/dL; 2 to < 6 years - 0.8 mg/dL; 6 to < 10 years- 1 mg/dL; 10 to < 13 years- 1.2 mg/dL; 13 to 15 years- 1.5 mg/dL for boys and 1.4 mg/dL for girls.

   OR

   Creatinine clearance or radioisotope GFR greater than or equal to 70ml/min/1.73 m2
9. Adequate Liver Function Defined As:

   * Bilirubin (sum of conjugated + unconjugated) less than or equal to 1.5 x upper limit of normal (ULN) for age
   * SGPT (ALT) less than or equal to 5 x upper limit of normal (ULN) for age
   * Serum albumin greater than or equal to 2 g/dL
10. Informed Consent: All patients and/or their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
11. Patients of child-bearing potential must have a negative pregnancy test and agree to use an effective birth control method (abstinence is an acceptable form of birth control).

Exclusion Criteria:

1. Extra-ocular retinoblastoma or retinoblastoma involving the anterior chamber
2. Retinoblastoma that could otherwise be treated with laser therapy, cryotherapy, or plaque therapy only
3. Structural brain abnormality
4. Uncontrolled infection, defined as requiring intravenous antibiotics at the time of enrollment
5. Concomitant Medications

   * Growth factors that support platelet or white cell number or function must not have been administered within 3 days prior to enrollment.
   * Patients who are currently receiving non-FDA approved drugs, or who have received a non-FDA approved drug within 7 days prior to enrollment, are ineligible.
   * Patients who are currently receiving other anti-cancer agents are ineligible.
6. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2011-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
1-year event-free survival (event defined as the need for external beam radiation or enucleation) | 1 year
Response rate of retinoblastoma to topotecan when administered directly into the ophthalmic artery. | Up to 18 weeks
  EUA and retCAM imaging will be used to assess response rate.
Local (ocular) toxicities associated with the proposed regimen. Toxicities assessed using clinical examinations (EUA and Teller cards and Allan figures or Snellen visual acuity charts or other measures as appropriate for child's age.) | Up to 12 months
  1. For non-verbal infants we will employ Teller cards or Reacts to Light (if vision is too poor for Teller cards)
  2. For pre-school age verbal toddlers/children we will employ LEA Symbols or HOTV, and possibly Allen figures
  3. For older children capable of reading an alphabet we will employ Snellen visual acuity charts. Standard methods to assess color vision will also be employed when feasible.
Patterns of response of retinoblastoma to topotecan when administered directly into the ophthalmic artery. | Up to 18 weeks
  Physical examination of the tumors will be recorded at baseline and at every tumor assessment visit. Tumors will be classified as having Type I, II, III, IV, V or O response based on characteristic features identified during physical examination.

SECONDARY OUTCOMES:
Visual pathway function | Up to 12 months
  Evaluation of visual pathway function will be measured using visual acuity, electroretinogram, visual evoked potential, and functional magnetic resonance imaging.
Pharmacokinetics (Cmax and AUC) of topotecan when administered directly into the ophthalmic artery. | Samples taken 15 and 60 minutes after topotecan administration on Day 1 of Cycle 1 (optional for patients)
Histologic findings in the eyes ultimately requiring enucleation. | At time of enucleation, only if indicated
  Any eye requiring enucleation will be assessed for the presence or absence of 'high risk' features defined as scleral or massive choroidal invasion of viable tumor, anterior chamber involvement, invasion of the optic nerve posterior to the lamina cribrosa, ciliary body or iris invasion.

CONTACTS AND LOCATIONS:
Overall Officials: James Geller, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Abruzzo TA, Geller JI, Kimbrough DA, Michaels S, Correa ZM, Cornell K, Augsburger JJ. Adjunctive techniques for optimization of ocular hemodynamics in children undergoing ophthalmic artery infusion chemotherapy. J Neurointerv Surg. 2015 Oct;7(10):770-6. doi: 10.1136/neurintsurg-2014-011295. Epub 2014 Sep 1. PMID 25179634